CLINICAL TRIAL: NCT04087460
Title: A Phase Ⅰa Randomized,Double-Blind, Placebo-controlled Clinical Trial to Preliminary Evaluate the Safety and Immunogenicity of Protein Based Pneumococcal Vaccine（PBPV） in Healthy People Aged Between 18 and 49 Years Old
Brief Title: Phase Ⅰa Clinical Trial of a Pneumococcal Vaccine
Acronym: PⅠCTPV
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: CanSino Biologics Inc. (Industry)
Collaborators: Henan Center for Disease Control and Prevention (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CS-CTP-PBPV-Ⅰa
Record Dates: First submitted 2019-09-10; First posted 2019-09-12 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-10

CONDITIONS: Pneumonia; Respiratory Tract Diseases; Respiratory Tract Infections
Keywords: Vaccnie; PspA; Pneomolysin
MeSH Terms: conditions — Pneumonia; Respiratory Tract Diseases; Respiratory Tract Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Low-dose Group A (Experimental): Subjects received three doses of PBPV with 20μg each antigen
  Interventions: Biological: Protein based pneumococcal vaccine(Low dose)
- Low-dose Group B (Placebo Comparator): Subjects received three doses of placebo
  Interventions: Biological: Protein based pneumococcal vaccine placebo(Low dose)
- Middle-dose Group A (Experimental): Subjects received three doses of PBPV with 50μg each antigen
  Interventions: Biological: Protein based pneumococcal vaccine(Middle dose)
- Middle-dose Group B (Placebo Comparator): Subjects received three doses of placebo
  Interventions: Biological: Protein based pneumococcal vaccine placebo(Middle dose)
- High-dose Group A (Experimental): Subjects received three doses of PBPV with 100μg each antigen
  Interventions: Biological: Protein based pneumococcal vaccine(High dose)
- High-dose Group B (Placebo Comparator): Subjects received three doses of placebo
  Interventions: Biological: Protein based pneumococcal vaccine placebo(High dose)

INTERVENTIONS:
Biological: Protein based pneumococcal vaccine(Low dose) — 0.2mL,Intramuscular other name:PBPV
  Arms: Low-dose Group A
Biological: Protein based pneumococcal vaccine placebo(Low dose) — 0.2mL,Intramuscular other name:PBPV placebo
  Arms: Low-dose Group B
Biological: Protein based pneumococcal vaccine(Middle dose) — 0.5mL,Intramuscular other name:PBPV
  Arms: Middle-dose Group A
Biological: Protein based pneumococcal vaccine placebo(Middle dose) — 0.5mL,Intramuscular other name:PBPV placebo
  Arms: Middle-dose Group B
Biological: Protein based pneumococcal vaccine(High dose) — 1.0mL,Intramuscular other name:PBPV
  Arms: High-dose Group A
Biological: Protein based pneumococcal vaccine placebo(High dose) — 1.0mL,Intramuscular other name:PBPV placebo
  Arms: High-dose Group B

SUMMARY:
Infections with Streptococcus pneumoniae often cause serious health problems, especially for infants and the elderly.Failure to cover all polysaccharide types is an even greater problem with adults than with children.

The aim of the study is to preliminary evaluate the safety and immunogenicity of PBPV vaccine compared to placebo,in order to provide a basis for subsequent clinical trial design.

DETAILED DESCRIPTION:
The polysaccharide vaccine protected 60% of elderly adults who were at risk for pneumococcal infection.However, pneumococci are highly diverse with respect to their capsular types , and the polysaccharide-protein conjugate vaccines will not protect against strains of the many capsular types not included in the vaccine.This experimental vaccine was covered 70% of all pneumococcal types, Subjects will receive three doses of PBPV vaccine on day 0,60 and 120 with different contents of 20μg,50μg,100μg each antigen in 18 to 49 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers aged 18 to 49 years old;
* Willing to provide proof of identity;
* Able to understand and sign the informed consent;
* Able and willing comply with the requirements of the protocol

Exclusion Criteria:

* Hypertensive volunteers with uncontrollable medications (on-site measurement: systolic blood pressure > 140 mmHg, diastolic blood pressure > 90 mmHg);
* Abnormal changes of laboratory measures (with clinical significance);
* Woman is pregnant and lactating (by urine pregnancy test)
* Suffered from pneumonia in the past three years;
* Invasive diseases caused by Streptococcus pneumoniae (such as meningitis, bacteremia, pericarditis, peritonitis, etc.) in the past three years;
* Allergic person;
* Any prior administration of blood products in last 3 month;
* Any prior administration of other research medicines in last 1 month;
* Plans to participate in or is participating in any other drug clinical study;
* Any prior administration of attenuated live vaccine in last 14 days;
* Any prior administration of subunit or inactivated vaccines in last 7 days;
* Had fever before vaccination, volunteers with temperature >37.0℃ on axillary setting;
* According to the investigator's judgment, the volunteers have any otherfactors that make them unfit to participate in the clinical trial

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2020-04-10 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Safety indexes of solicited and unsolicited adverse reactions | within 30 minutes,0-7 days,0-30 days post-vaccination
  Occurrence of solicited and unsolicited reactions post each vaccination
Safety indexes of lab measures | day 3 and 8 post the first vaccination
  Occurrence of abnormal changes of hematological examination,clinical chemistry test,urine test and vital signs
Safety indexes of lab measures | day 14 and 30 post each vaccination
  Occurrence of abnormal changes of CK-MB,CTN,urine test and vital signs

SECONDARY OUTCOMES:
safety indexes of SAE | within 180 days post vaccination
  Occurrence of SAE
immunogencity indexes of GMC and GMI by ELISA | day 8, 14,30,60 post each vaccination
  Geometric mean concentration(GMC) and Geometric mean increase（GMI）of anti-PspA-RX1 , anti-PspA-3296, anti-PspA-5668 and anti-PlyLD antibodies in serum
immunogencity indexes of the seropositivity rates by ELISA | day 8, 14,30,60 post each vaccination
  the seropositivity rates of anti-PspA-RX1 , anti-PspA-3296, anti-PspA-5668 and anti-PlyLD antibodies in serum

OTHER OUTCOMES:
immunogencity indexes of GMT and GMI by Opsonophagocytic assay (OPA) | day30,60 post each vaccination
  Geometric mean titer(GMT) and Geometric mean increase（GMI）of antibodies in serum
immunogencity indexes of neutralization test | day30,60 post each vaccination
  neutralization test activity of anti-Ply antibody in serum

CONTACTS AND LOCATIONS:
Overall Officials: Xia Shengli, Principal Investigator — Henan Province Center for Disease Control and Prevention
Locations (1):
- Suixian Center for Disease Control and Prevention, Shangqiu, Henan, China

IPD SHARING:
Plan to Share IPD: No
In order to maintain the rights of the subject, do not open the IPD